CLINICAL TRIAL: NCT02695563
Title: Influence of Vaginal Lactoferrin Administration Prior to Genetic Amniocentesis on PGE2, MMP-9, MMP-2, TIMP-1 and TIMP-2 Amniotic Fluid Concentrations
Brief Title: Effects of Vaginal Lactoferrin Administration Prior to Genetic Amniocentesis on Inflammatory Mediators
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Università degli Studi di Ferrara (Other)
Responsible Party: Principal Investigator, Alessandro Trentini, PhD, Università degli Studi di Ferrara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRUa1GR-2013-00000220
Record Dates: First submitted 2016-02-24; First posted 2016-03-01 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-03

CONDITIONS: Pregnancy
Keywords: Amniocentesis
MeSH Terms: interventions — Lactoferrin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- controls (No Intervention): The patients will be not treated with vaginal lactoferrin
- Lactoferrin (Active Comparator): The patients will be administered with a single dose of 300 mg vaginal lactoferrin 4 hours prior to mid-trimester genetic amniocentesis.
  Interventions: Drug: Lactoferrin

INTERVENTIONS:
Drug: Lactoferrin
  Arms: Lactoferrin

SUMMARY:
The aim of the study is to evaluate the effect of vaginal lactoferrin administration on amniotic fluid PGE2 level and MMP-TIMP system in women undergoing genetic amniocentesis. Two groups of patients will be prospectively enrolled: not treated with lactoferrin and treated with vaginal lactoferrin 4 hours prior to mid-trimester genetic amniocentesis.

DETAILED DESCRIPTION:
Pregnant women undergoing genetic amniocentesis within the 16th-18th gestational week will be enrolled at the Obstetric Unit, University of Ferrara.

The selected patients will be randomly assigned to receive a vaginal compound containing 300 mg of lactoferrin 4 hours before amniocentesis or they will be untreated (controls).

Amniotic fluid samples will be obtained by transabdominal amniocentesis and the sample not required for clinical purposes will be centrifuged to remove particulate material and the supernatants will be aliquoted and stored at -80°C until assay.

ELIGIBILITY:
Inclusion Criteria:

* singleton gestation
* maternal age as indication to fetal karyotyping

Exclusion Criteria:

* consumption of drugs interfering with the immune system
* previous miscarriages
* pregnancy at risk for maternal or fetal disease
* lactose intolerance

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 111 (Actual)
Dates: Start 2014-01; Primary Completion 2015-03 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Measurement of inflammatory markers in the amniotic fluid | 1 month after the enrollment of patients will be concluded.
  The investigator will measure the amniotic fluid concentration of Prostaglandin E2(PGE2), active MMP(Matrix Metalloproteinase)-9, active MMP-2, TIMP(Tissue Inhibitor of Matrix Metalloproteinase)-1 and TIMP-2 by commercially available ELISA or activity assay systems; concentration of creatinine in the amniotic fluids will be measured by the alkaline picrate method. Controls and Lactoferrin-treated patients will be compared by parametric or non-parametric statistical tests.

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Contini, Professor, Study Director — Section of Dermatology and Infectious Diseases, Department of Medical Sciences, University of Ferrara
Locations (1):
- Obstetric Unit, University of Ferrara, Cona, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Trentini A, Maritati M, Rosta V, Cervellati C, Manfrinato MC, Hanau S, Greco P, Bonaccorsi G, Bellini T, Contini C. Vaginal Lactoferrin Administration Decreases Oxidative Stress in the Amniotic Fluid of Pregnant Women: An Open-Label Randomized Pilot Study. Front Med (Lausanne). 2020 Sep 8;7:555. doi: 10.3389/fmed.2020.00555. eCollection 2020. PMID 33015104
- [Derived] Trentini A, Maritati M, Cervellati C, Manfrinato MC, Gonelli A, Volta CA, Vesce F, Greco P, Dallocchio F, Bellini T, Contini C. Vaginal Lactoferrin Modulates PGE2, MMP-9, MMP-2, and TIMP-1 Amniotic Fluid Concentrations. Mediators Inflamm. 2016;2016:3648719. doi: 10.1155/2016/3648719. Epub 2016 Oct 31. PMID 27872513